CLINICAL TRIAL: NCT01075087
Title: TAP) Block in Morbid Obese Patients Undergoing Laparoscopic Gastric Bypass Surgery: A Prospective,Randomized, Blinded Study
Brief Title: The Effect of Pre-Operative Transversus Abdominis Plane (TAP) Block in the Post Operative Opioid Consumption in Morbid Obese Patients Undergoing Laparoscopic Gastric Bypass Surgery: A Prospective,Randomized, Blinded Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00023482
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-05

CONDITIONS: Pain; Obesity; Surgery
Keywords: TAP Block; Pain; Obesity; Surgery; Laparoscopic Banding
MeSH Terms: conditions — Pain; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): (control group) will receive sterile normal saline in the block
  Interventions: Drug: Placebo
- Active comparator (Active Comparator): (study group) will receive a bilateral TAP block using 20 cc of 0.5% ropivacaine on each side.
  Interventions: Drug: (study group) will receive a bilateral TAP block using 20 cc of 0.5% ropivacaine on each side.

INTERVENTIONS:
Drug: Placebo — Bilateral TAP block using sterile normal saline.
  Arms: Placebo
Drug: (study group) will receive a bilateral TAP block using 20 cc of 0.5% ropivacaine on each side. — (study group) will receive a bilateral TAP block using 20 cc of 0.5% ropivacaine on each side.
  Arms: Active comparator

SUMMARY:
The use of preoperative TAP block in laparoscopic bariatric surgery can improve the postoperative pain and quality of recovery in patients undergoing these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* BMI >35 Kg/m2
* Surgery: laparoscopic gastric bypass surgery
* ASA status: I, II and III
* Fluent in English

Exclusion Criteria:

* History of allergy to local anesthetics
* Chronic opioid use
* Pregnant patients
* Patients who remained intubated after surgery

Drop-out criteria:

Patient or surgeon request Complications related to the procedure or conversion to open route Patient requiring mechanical ventilation after surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio DeOliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Mun EC, Blackburn GL, Matthews JB. Current status of medical and surgical therapy for obesity. Gastroenterology. 2001 Feb;120(3):669-81. doi: 10.1053/gast.2001.22430. PMID 11179243
- [Background] Peiser J, Lavie P, Ovnat A, Charuzi I. Sleep apnea syndrome in the morbidly obese as an indication for weight reduction surgery. Ann Surg. 1984 Jan;199(1):112-5. doi: 10.1097/00000658-198401000-00020. PMID 6691724
- [Background] Kyzer S, Charuzi I. Obstructive sleep apnea in the obese. World J Surg. 1998 Sep;22(9):998-1001. doi: 10.1007/s002689900506. PMID 9717428
- [Background] Rosenberg-Adamsen S, Kehlet H, Dodds C, Rosenberg J. Postoperative sleep disturbances: mechanisms and clinical implications. Br J Anaesth. 1996 Apr;76(4):552-9. doi: 10.1093/bja/76.4.552. No abstract available. PMID 8652329
- [Background] Alexander CM, Gross JB. Sedative doses of midazolam depress hypoxic ventilatory responses in humans. Anesth Analg. 1988 Apr;67(4):377-82. PMID 3354874
- [Background] Dhonneur G, Combes X, Leroux B, Duvaldestin P. Postoperative obstructive apnea. Anesth Analg. 1999 Sep;89(3):762-7. doi: 10.1097/00000539-199909000-00045. PMID 10475322
- [Background] Chung F, Crago RR. Sleep apnoea syndrome and anaesthesia. Can Anaesth Soc J. 1982 Sep;29(5):439-45. doi: 10.1007/BF03009406. PMID 6751498
- [Background] Passannante AN, Tielborg M. Anesthetic management of patients with obesity with and without sleep apnea. Clin Chest Med. 2009 Sep;30(3):569-79, x. doi: 10.1016/j.ccm.2009.05.009. PMID 19700053
- [Background] Wills VL, Hunt DR. Pain after laparoscopic cholecystectomy. Br J Surg. 2000 Mar;87(3):273-84. doi: 10.1046/j.1365-2168.2000.01374.x. PMID 10718794
- [Background] Goldstein A, Grimault P, Henique A, Keller M, Fortin A, Darai E. Preventing postoperative pain by local anesthetic instillation after laparoscopic gynecologic surgery: a placebo-controlled comparison of bupivacaine and ropivacaine. Anesth Analg. 2000 Aug;91(2):403-7. doi: 10.1097/00000539-200008000-00032. PMID 10910857
- [Background] Shaw IC, Stevens J, Krishnamurthy S. The influence of intraperitoneal bupivacaine on pain following major laparoscopic gynaecological procedures. Anaesthesia. 2001 Nov;56(11):1041-4. doi: 10.1046/j.1365-2044.2001.02215.x. PMID 11703235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled consecutively from 03/2010 through 07/2012 in the pre operative area of the hospital.
Pre-assignment Details: 26 were assessed for eligibility. 7 were excluded ( 4 did not meet inclusion criteria and 3 refused to participate).
Period: Overall Study
Arm/Group | Placebo | Active Comparator
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active Comparator | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Median (Full Range); unit: years] | 50 [36 to 54] | 47 [39 to 53] | 48 [36 to 54]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery 40 Score
Description: Quality of Recovery 40 Score at 24 hours postoperative.
Time Frame: 24 hours post operatively
Measure: Median (Inter-Quartile Range); unit: units on scale 40 (low) - 200 (high)
Arm/Group | Placebo | Active Comparator
Number analyzed (Participants) | 9 | 10
units on scale 40 (low) - 200 (high) | 170 [160 to 175] | 175.5 [170 to 189]
Statistical Analysis 1: Comparison: Placebo vs Active Comparator; Test type: Superiority or Other; p = .05, Wilcoxon (Mann-Whitney); Median Difference (Net) = -5.5, 90% CI 2-sided [-26 to 3]

2. Secondary Outcome: 24 Hour Total Opioid Consumption.
Description: 24 Hour total opioid consumption translated into IV morphine equivalents.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: miligram IV morphine equivalents
Arm/Group | Placebo | Active Comparator
Number analyzed (Participants) | 9 | 10
miligram IV morphine equivalents | 13 [7 to 21.5] | 7.5 [2.5 to 11.5]

ADVERSE EVENTS:
Arm/Group | Placebo | Active Comparator
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 3/9 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Active Comparator (N=10)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes